CLINICAL TRIAL: NCT04242901
Title: Serial Faecal Immunochemical Testing in Patients With Colorectal Cancer
Brief Title: 4-week Serial FIT Analysis in Patients With CRC
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19ON031
Record Dates: First submitted 2020-01-09; First posted 2020-01-27 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
Keywords: FIT; Symptomatic FIT
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer: Patients recently diagnosed colorectal cancer
  Interventions: Diagnostic Test: Faecal Immunochemical Test - OC Sensor, Eiken, Tokyo

INTERVENTIONS:
Diagnostic Test: Faecal Immunochemical Test - OC Sensor, Eiken, Tokyo — Quantitative Faecal Immunochemical Test - OC Sensor, Eiken, Tokyo

SUMMARY:
Assimilation of FIT into primary and secondary care diagnostic pathways will lead to an increased prominence of the investigation in the diagnosis of colorectal cancer (CRC). Questions remain about whether serial FIT analysis improves accuracy, and what factors affect it.

Our study will analyse FIT results in recently diagnosed CRC patients to determine the risk of a false-negative FIT result and evaluate whether repeated analysis improves diagnostic accuracy. The study aims to advise on whether there is an optimal interval between sample collection to improve diagnostic accuracy and whether any patients are at risk of a false negative based on demographics, medications or other pathological factors.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) remains a leading cause of cancer death in the UK and worldwide. Improving outcomes depends in part on achieving earlier diagnosis of the disease.

The Faecal Immunochemical Test (FIT) is replacing the less accurate Faecal Occult Blood Test (FOBT) in the UK and has the potential to help achieve earlier stage diagnosis of CRC. Whilst FIT has been validated as a screening test for the Bowel Cancer Screening Programme (BCSP), its role in diagnosing CRC in symptomatic populations is yet to be defined.

Nottingham is a pioneering centre using FIT to stratify risk and determine first-investigation in its two-week-wait (2WW) pathway. To optimise use of FIT and minimise the chance of missed cancers, this project aims to better understand variation of FIT results over time and how certain factors affect FIT result.

Much of the literature has focused on the evaluation of FIT in an asymptomatic population, which is inherently low risk (4,6,7). Expanding use of FIT to stratify risk and guide investigations for cancer in (higher risk) symptomatic populations necessitates a thoroughly evaluated testing strategy. At present there is insufficient information to advise on "negative" FIT results in symptomatic patients. This study will comprehensively measure FIT variation over time in patients with the target condition (CRC) and help answer whether additional samples are likely to improve accuracy of FIT.

Risk factors for false positives and false negatives have been previously identified but are not widely established (4). Our study will record the presence of these risk factors, and evaluate their effects on FIT-positivity with subsequent statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer

Exclusion Criteria:

* Less than 18 years old
* Not attending Nottingham University Hospitals for diagnosis/treatment (attending another trust)
* No histological diagnosis of colorectal cancer
* Unable to provide informed consent - for example due to language barriers or lacking capacity to join study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients will be recruited to the study. Nottingham University Hospitals NHS Trust diagnoses approximately 500 CRCs per year, yielding an available population pool of 1000 patients in the study period. A sample size of 200 participants (returning 1000 samples in total) represents a realistic recruitment target.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
False negative FIT results - Determine the occurrence of falsely negative FIT results in the presence of colorectal cancer | 2 years
  Determine the occurrence of falsely negative FIT results in the presence of colorectal cancer
Number of participants who yield sequential FIT results in divergent strata used for clinical decision making | 2 years
  Number of participants who yield sequential FIT results in divergent strata used for clinical decision making (FIT <4 μg Hb/g faeces, 4-9.9 μg Hb/g faeces, 10-99.9 μg Hb/g faeces, 100-150 μg Hb/g faeces, >150 μg Hb/g faeces)

SECONDARY OUTCOMES:
Calculation of Odds Ratios for age, gender, family history of CRC, hypertension, obesity, smoking status, excessive alcohol intake, right sided tumour, stage 1 cancer | 2 years
  Calculation of Odds Ratios for age, gender, family history of CRC, hypertension, obesity, smoking status, excessive alcohol intake, right sided tumour, stage 1 cancer

CONTACTS AND LOCATIONS:
Overall Officials: David Humes, MBBS, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data